CLINICAL TRIAL: NCT01101438
Title: A Phase III Randomized Trial of Metformin Versus Placebo on Recurrence and Survival in Early Stage Breast Cancer
Brief Title: A Phase III Randomized Trial of Metformin vs Placebo in Early Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); ETOP IBCSG Partners Foundation (Network); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA32; U10CA077202 (NIH); CAN-NCIC-MA.32 (Other: PDQ Identifier); CDR0000669788 (Other: PDQ)
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIC breast cancer; male breast cancer; HER2-negative breast cancer; estrogen receptor-positive breast cancer; HER2-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral metformin hydrochloride twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in receptor positive (ER and/or PgR positive) subjects in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: metformin hydrochloride
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in receptor positive (ER and/or PgR positive) subjects in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: metformin hydrochloride — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
This study is looking at whether Metformin, an agent that is commonly used to treat diabetes, can decrease or affect the ability of breast cancer cells to grow and whether Metformin will work with other therapies to keep cancer from recurring. Health Canada has not approved the sale or use of Metformin to treat breast cancer, although they have approved its use in this clinical trial. Although Metformin is approved by the FDA for the treatment of diabetes, its use in breast cancer is considered investigational.

DETAILED DESCRIPTION:
This is a multicenter study. Patients are stratified according to hormone-receptor status (estrogen receptor- and/or progesterone receptor- positive vs both receptors negative), body mass index (≤ 30 vs > 30 kg/m²), HER2 status (positive vs negative), and prior chemotherapy (any vs none). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral metformin hydrochloride twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in the absence of disease progression or unacceptable toxicity.

Blood and tumor samples are collected periodically for correlative studies.

Patients may complete quality-of-life, physical activity, and diet questionnaires at baseline and at 6, 12, 24, 36, 48, and 60 months. (Sub-set of patients).

After completion of study treatment, patients are followed annually.

ELIGIBILITY:
Eligibility Criteria:

* Subjects must have histologically confirmed invasive breast cancer and be enrolled in the trial within 12 months after the first histologic diagnosis of invasive breast cancer. A core biopsy interpreted as invasive cancer meets this criterion; otherwise, the date of first histologic diagnosis will be the date of first surgical procedure that identifies invasive cancer (biopsy, lumpectomy or mastectomy). Neoadjuvant subjects should have no evidence of clinical T4 disease prior to chemotherapy and surgery. Bilateral breast carcinoma is allowed provided diagnoses are synchronous - that is, within 3 months of one another - and at least one of the two breast carcinomas meet the eligibility criteria and neither violates the eligibility criteria.
* All subjects (both adjuvant and neo-adjuvant) must have sentinel lymph node biopsy and/or axillary lymph node dissection.

Sentinel lymph node biopsy alone is allowed in the following instances:

1. sentinel lymph node biopsy is negative: pN0
2. sentinel lymph node biopsy is positive for isolated tumour cells only: pN0 (i+)
3. * clinically node negative, T1-2 tumours with sentinel lymph node biopsy positive in ≤ 2 lymph nodes without extra-capsular extension or matted nodes and undergoing breast conserving surgery and tangential whole breast irradiation (* excludes subjects treated with neo-adjuvant systemic therapy)

Definitive surgery and/or chemotherapy have been completed at least 4 weeks prior to randomization. Surgical margins must be clear of invasive carcinoma. If there is microscopic residual ductal in situ disease present at lumpectomy or total mastectomy margins, further excision is highly recommended. If further excision is not undertaken, the subject may still be entered on study, provided that in addition to breast or chest wall irradiation, a boost to the tumour bed is delivered. In situ lobular disease at the margin is acceptable.

Adjuvant subjects with the following pT pN combinations are eligible:

* pT1c, pN0 AND negative estrogen and progesterone receptors AND HER2 negative OR
* pT2N0 and at least one of the following tumour characteristics: histologic grade 3, lymphovascular invasion, negative estrogen and progesterone receptors, HER2 positive, Oncotype Dx recurrence score ≥ 25 (or if Oncotype Dx recurrence score is not available, Ki67 > 14%) OR
* Subjects with pT3, pN0 OR
* Subjects with pT1-3, pN1-3

The eligibility of neo-adjuvant subjects is assessed on the basis of cTNM. The same eligible TNM combinations apply.

* HER2 status must be known. (Positive = 3+ over-expression by IHC in > 30% of invasive tumour cells OR HER2 gene amplification by FISH/CISH > 6 HER2 gene copies per nucleus, OR a FISH/CISH ratio: HER2 gene copies to chromosome 17 signals of ≥ 2.2. All other results will be considered negative).
* Patients must have had a bilateral mammogram within 12 months prior to randomization, unless the initial surgery was a total mastectomy, in which case only a mammogram of the remaining breast is required. (Subjects with bilateral total mastectomies and no mammogram within 12 months prior to randomization must, instead, have a physical examination of the chest wall to ensure there is no residual or recurrent disease at the time of randomization. The date of this examination is used in place of the mammogram date on the eligibility checklist.)
* Investigations, including chest X-ray or CT chest, bone scan (with radiographs of suspicious areas) and abdominal ultrasound or liver scan or CT abdomen have been performed between the first histologic diagnosis and the time of randomization.

  * Chest X-Ray, 2 view (or Chest CT) is mandatory
  * Bone scans (with x-rays of abnormal areas) are required only if there are signs or symptoms of metastatic disease
  * Abdominal imaging is required only if there are signs or symptoms of metastatic disease
* Hematology investigations (WBC, Granulocytes, Platelets, Hemoglobin) have been completed within 28 days prior to randomization and results are available.
* Biochemistry investigations have been completed within 28 days prior to randomization and values are within the parameters required by the protocol.

AST < 1.8 X ULN; ALT < 1.8 X ULN; Alkaline Phosphatase < 2 X ULN; Serum Creatinine < 115 μmol/L (1.3mg/dL) Serum Bilirubin < institution ULN (except for subjects with Gilbert's Disease who are eligible despite elevated serum bilirubin level)

* ECOG Performance Status of 0,1 or 2 (at baseline evaluation visit within 28 days prior to randomization).
* Age ≥ 18 and < 75 and life expectancy of at least 5 years (18 years of age was used as a cut-off due to the lack of data indicating that breast cancer is a health issue in the < 18 years age group and metformin safety in pediatric patients has not been confirmed. Age > 80 carries increased risk of lactic acidosis and study intervention is for 5 years).
* Subjects must be accessible for treatment and follow-up. Investigators must assure themselves the subjects randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 10 working days of patient randomization.
* Subject consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is given. A copy of the initial full board REB approval and approved consent form must be sent to the central office. The patient must sign the consent form prior to randomization or registration. Please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records (see Section 16 for further details).

For the first 888 eligible English or French-speaking subjects only (sub-set enrollment completed 2011NOV04):

* Subject is able (i.e. sufficiently fluent) and willing to complete the Quality of Life (EORTC QLQ C-30 and Trial Specific Checklist) in English or French. The baseline assessment must already have been completed at the time of enrollment. Inability (illiteracy in English or French, loss of sight or other equivalent reason) to complete questionnaires will not make the patient ineligible for the study; however, ability but unwillingness to complete the questionnaires will make the patient ineligible. (Once the target number of 888 subjects is achieved, this criterion will no longer need to be fulfilled.) [See Appendix VI]. Sub-set enrollment completed 2011NOV04.
* English-speaking subjects who have completed the Quality of Life Questionnaire who are able (i.e. sufficiently fluent) and willing to complete Nurses Health Study II Physical Activity Questionnaire and Block Alive Screener in English. The baseline assessment must already have been completed at the time of enrollment. Inability (illiteracy in English, loss of sight or other equivalent reason) to complete questionnaires will not make the patient ineligible for the study; however, ability but unwillingness to complete the questionnaires will make the patient ineligible. (This component of the study will close at the same time as the Quality Of Life sub-study.) Closed to new patient enrollment as of 2011NOV04.

Ineligibility Criteria:

* Subjects with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Subjects with locally recurrent or metastatic breast carcinoma. (Subjects with prior invasive breast cancer at any time are not eligible. Subjects with prior DCIS only in either breast are eligible provided the DCIS has been curatively treated including surgery, radiotherapy and/or Tamoxifen).
* Subjects whose axillary node status is unknown.
* Known diabetes (type 1 or 2) or baseline fasting glucose > 7.0 mmol/L (126 mg/dL). (Sampled and assayed according to local institution's procedures.)
* Known hypersensitivity or intolerance to metformin.
* Any condition associated with increased risk of metformin-associated lactic acidosis (e.g. congestive heart failure defined as New York Heart Association {NYHA} Class III or IV functional status [see Appendix IX], history of acidosis of any type; habitual * Currently taking metformin, sulfonylureas, thiazolidinediones or insulin for any reason.
* Current or planned pregnancy or lactation in women of child-bearing potential. Men should not father a child. (An effective method of birth control should be used while on study treatment which could include abstinence, IUD, condoms or other barrier methods of birth control because the safety of metformin in pregnancy or in male fertility has not been established).
* Concurrent or planned participation in randomized trials of weight loss or exercise interventions or trials targeting insulin, IGF-1 or their receptors, or involving P13K inhibitors (at the time of randomization)*.
* These interventions would interfere with the primary endpoint. (Also, in general, double randomizations in breast cancer trials for MA.32 patients are permitted only if the patient meets all the eligibility criteria for MA.32 and the sponsor of the previous trial has no objection to the patient also being enrolled in MA.32).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3649 (Actual)
Dates: Start 2010-08-13 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J. Goodwin, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (344):
- United States (280):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Pinnacle Oncology Associates, Scottsdale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Cancer Center at University Medical Center North, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Enloe Medical Center, Chico, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Kaiser Permanente, Hayward, Hayward, California
  - Moores University of California San Diego Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - University of Southern California, Los Angeles, California
  - University of California at Los Angeles (UCLA ), Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Bay Area Tumor Institution CCOP, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis-Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-Mission, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - University of California San Francisco Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Stanford University, Stanford, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center, Walnut Creek, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Connecticut Oncology and Hematology LLP, Torrington, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - Mount Sinai Medical Center CCOP, Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Rush - Copley Medical Center, Aurora, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Resurrection Healthcare, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Foundation - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Indiana University Hospital/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Howard Regional Healthcare System, Kokomo, Indiana
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - McFarland Clinic, Ames, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Kansas City CCOP, Prairie Village, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Owensboro Mercy Medical Center, Owensboro, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - York Hospital, York Village, Maine
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Saint Vincent Hospital - Fallon Clinic, Worcester, Massachusetts
  - University of Michigan Health System-Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System, Battle Creek, Michigan
  - Wayne State University, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Health Partners-Mercy Campus, Muskegon, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic CCOP, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Saint John's Hospital, Springfield, Missouri
  - Cox Medical Center, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Good Samaritan Hospital, Kearney, Nebraska
  - Lincoln Medical Education Foundation Cancer Resource Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium CCOP, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - New Hampshire Oncology-Hematology PA, Concord, New Hampshire
  - New Hampshire Oncology Hematology Associates, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York PC, East Syracuse, New York
  - Monter Cancer Center, Lake Success, New York
  - North Shore University Hospital CCOP, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Kisco Medical Group at Northern Westchester Hospital, Mount Kisco, New York
  - Mount Kisco Medical Group, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Saint Luke's Roosevelt Hospital Center - Saint Luke's Division, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - The North Division of Montefiore Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Forsyth Memorial Hospital, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Medcenter One Health Systems, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Columbia River Oncology Program, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Saint Joseph Medical Center, Reading, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University Medical Center Brackenridge, Austin, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Saint John Medical Center, Longview, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Rockwood Clinic, Spokane, Washington
  - Northwest CCOP, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program, Fond du Lac, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Health System/CCOP, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Wheaton Franciscan Healthcare - Saint Joseph, Milwaukee, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
- Canada (41):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Centre - West Toronto, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUM - Hotel Dieu du Montreal, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Switzerland (8):
  - Switzerland-Chur (Ratisches Kantons- und Regionalspital), Chur
  - Brustzentrum Thurgau, Spital Thurgau AG, Frauenfeld
  - Fondazione Oncologia Lago Maggiore, FOLM, Locarno
  - Switzerland-Luzern (Kantonsspital Luzern), Lucerne
  - Switzerland - Oncology Institute of Southern Switzerland (IOSI), Mendrisio
  - Switzerland - Olten (Kantonsspital) affiliate-3101, Olten
  - Switzerland - ZeTup St.Gallen, Sankt Gallen
  - Switzerland - Brust-Zentrum, Zurich, Zurich
- United Kingdom (15):
  - University Hospital Birmingham NHS Foundation Trust, Edgbaston, Birmingham
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh, Crewe Road South
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Medway NHS Foundation Trust, Gillingham, Kent
  - Kent Centre for Oncology, Maidstone, Kent
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough, Marton Road
  - Withybush General Hospital, Haverfordwest, Pembrokeshire
  - East and North Hertfordshire NHS Trust, Middlesex, Rickmansworth Road
  - Singleton Hospital, Swansea, Sketty Lane
  - North Bristol NHS Trust, Bristol, Southmead
  - St George's Healthcare NHS Trust, London, Tooting
  - Ninewells Hospital, Dundee, University of Dundee
  - Velindre Cancer Centre, Cardiff, Whitchurch
  - The Christie NHS Foundation Trust, Manchester, Withington
  - Sandwell and West Birmingham Hospitals NHS Trust, Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodwin PJ, Parulekar WR, Gelmon KA, Shepherd LE, Ligibel JA, Hershman DL, Rastogi P, Mayer IA, Hobday TJ, Lemieux J, Thompson AM, Pritchard KI, Whelan TJ, Mukherjee SD, Chalchal HI, Oja CD, Tonkin KS, Bernstein V, Chen BE, Stambolic V. Effect of metformin vs placebo on and metabolic factors in NCIC CTG MA.32. J Natl Cancer Inst. 2015 Mar 4;107(3):djv006. doi: 10.1093/jnci/djv006. Print 2015 Mar. PMID 25740979
- [Result] Goodwin PJ, Chen BE, Gelmon KA, Whelan TJ, Ennis M, Lemieux J, Ligibel JA, Hershman DL, Mayer IA, Hobday TJ, Bliss JM, Rastogi P, Rabaglio-Poretti M, Mukherjee SD, Mackey JR, Abramson VG, Oja C, Wesolowski R, Thompson AM, Rea DW, Stos PM, Shepherd LE, Stambolic V, Parulekar WR. Effect of Metformin vs Placebo on Invasive Disease-Free Survival in Patients With Breast Cancer: The MA.32 Randomized Clinical Trial. JAMA. 2022 May 24;327(20):1963-1973. doi: 10.1001/jama.2022.6147. PMID 35608580
- [Derived] Goodwin PJ, Chen BE, Gelmon KA, Whelan TJ, Ennis M, Lemieux J, Ligibel JA, Hershman DL, Mayer IA, Hobday TJ, Bliss JM, Rastogi P, Rabaglio-Poretti M, Thompson AM, Rea DW, Stos PM, Shepherd LE, Stambolic V, Parulekar WR. Effect of Metformin Versus Placebo on New Primary Cancers in Canadian Cancer Trials Group MA.32: A Secondary Analysis of a Phase III Randomized Double-Blind Trial in Early Breast Cancer. J Clin Oncol. 2023 Dec 10;41(35):5356-5362. doi: 10.1200/JCO.23.00296. Epub 2023 Sep 11. PMID 37695982

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Patients receive oral metformin hydrochloride (850mg) twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in receptor positive (ER and/or PgR positive) subjects in the absence of disease progression or unacceptable toxicity.
  metformin hydrochloride: Given orally
- Placebo: Patients receive oral placebo (850mg) twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in receptor positive (ER and/or PgR positive) subjects in the absence of disease progression or unacceptable toxicity.
  placebo: Given orally
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 1824 | 1825
Completed | 1816 | 1816
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 8 | 9

BASELINE CHARACTERISTICS:
Population: All randomized patients will be analyzed according to the arm that they were randomized to (intent to treat population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 1824 | 1825 | 3649
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.18 (10.05) | 52.56 (10.12) | 52.37 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1821 | 1822 | 3643
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 8 | 17
  Asian | 51 | 48 | 99
  Native Hawaiian or Other Pacific Islander | 5 | 8 | 13
  Black or African American | 83 | 84 | 167
  White | 1653 | 1651 | 3304
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 26 | 49
Region of Enrollment [Number; unit: participants]
  Canada | 599 | 604 | 1203
  United States | 1132 | 1127 | 2259
  United Kingdom | 68 | 69 | 137
  Switzerland | 25 | 25 | 50
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] | 28.72 (6.58) | 28.52 (6.22) | 28.62 (6.40)
Hormone Receptor [Count of Participants; unit: Participants] — Hormone receptor is a special protein that in a breast cancer cell that enables the cell to grow in the presence of estrogen or progesterone that is measured using standard methods in the laboratory where the diagnosis was made.
  Participants
    Positive | 1268 | 1265 | 2533
    Negative | 556 | 560 | 1116

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-free Survival in Hormone Receptor (ER and PgR) Positive Sub-groups
Description: Invasive disease-free survival (IDFS) is defined as percentage of patients without documented development of ipsilateral and contralateral invasive breast tumour, local/regional invasive recurrence, distant recurrence, death from any causes. If a subject has not had invasive disease or died at the time of data cut-off for this final analysis, IDFS was censored on the date of last follow-up.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients without event
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 1268 | 1265
percentage of patients without event | 86.5 [84.5 to 88.5] | 85.9 [83.9 to 87.9]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.93, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.84 to 1.21]

2. Primary Outcome: Invasive Disease-free Survival
Description: Invasive disease-free survival (IDFS) is defined as the percent of patients without documented development of ipsilateral and contralateral invasive breast tumour, local/regional invasive recurrence, distant recurrence, death from any causes. If a subject has not had invasive disease or died at the time of data cut-off for this final analysis, IDFS was censored on the date of last follow-up.
Time Frame: 5 years
Population: All randomized patients will be analyzed according to the arm that they were randomized to (intent to treat population).
Measure: Number (95% Confidence Interval); unit: percentage of patients without event
Groups:
- Metformin: Patients receive oral metformin hydrochloride twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in receptor positive (ER and/or PgR positive) subjects in the absence of disease progression or unacceptable toxicity.
  metformin hydrochloride: Given orally
- Placebo: Patients receive oral placebo twice daily (once daily in weeks 1-4). Treatment continues for up to 5 years in receptor positive (ER and/or PgR positive) subjects in the absence of disease progression or unacceptable toxicity.
  placebo: Given orally
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 1824 | 1825
percentage of patients without event | 84.9 [83.2 to 86.6] | 84.1 [82.4 to 85.8]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.94, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.87 to 1.17]

3. Secondary Outcome: Overall Survival
Description: Number of patients who died from any causes.
Time Frame: 10 years
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 1824 | 1825
Participants
  Patients who died | 201 | 198
  Patients who alive | 1623 | 1627
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.88, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.83 to 1.24]

4. Secondary Outcome: Distant Relapse-free Survival
Description: Distant Relapse Free Survival (DRFS) is defined as the percentage of patients without any documented distant recurrence, death from breast cancer, death from a non breast cancer cause or death from an unknown cause. If a subject has not had distant DRFS event nor died at the time of data cut-off for this analysis, DRFS will be censored on the date of last disease assessment.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients without event
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 1824 | 1825
percentage of patients without event | 88.7 [87.2 to 90.2] | 87.8 [86.3 to 89.3]

5. Secondary Outcome: Breast Cancer-specific Mortality
Description: Patients who died from breast cancer
Time Frame: 10 years
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 1824 | 1825
Participants | 155 | 160

ADVERSE EVENTS:
Time Frame: 10 years
Description: For all cause mortality, the analysis population is intent to treat, which includes all randomized patients. This is different from the analysis population for the adverse event and serious adverse event (treated population).
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 201/1824 | 198/1825
Serious Adverse Events (participants affected / at risk) | 1/1816 | 3/1816
Other Adverse Events (participants affected / at risk) | 1707/1816 | 1670/1816
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=1816) | Placebo (N=1816)
Retinal vascular disorder (Eye disorders) | 0 | 1
Fetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=1816) | Placebo (N=1816)
Abdominal pain (Gastrointestinal disorders) | 191 | 146
Bloating (Gastrointestinal disorders) | 179 | 151
Constipation (Gastrointestinal disorders) | 288 | 226
Diarrhea (Gastrointestinal disorders) | 819 | 354
Dyspepsia (Gastrointestinal disorders) | 174 | 141
Flatulence (Gastrointestinal disorders) | 155 | 145
Gastroesophageal reflux disease (Gastrointestinal disorders) | 121 | 114
Nausea (Gastrointestinal disorders) | 560 | 297
Vomiting (Gastrointestinal disorders) | 139 | 100
Edema limbs (General disorders) | 143 | 130
Fatigue (General disorders) | 811 | 797
Pain (General disorders) | 250 | 276
Dermatitis radiation (Injury, poisoning and procedural complications) | 127 | 138
Weight gain (Investigations) | 90 | 156
Weight loss (Investigations) | 171 | 81
Anorexia (Metabolism and nutrition disorders) | 182 | 84
Hyperglycemia (Metabolism and nutrition disorders) | 80 | 93
Arthralgia (Musculoskeletal and connective tissue disorders) | 389 | 427
Arthritis (Musculoskeletal and connective tissue disorders) | 86 | 99
Back pain (Musculoskeletal and connective tissue disorders) | 211 | 189
Bone pain (Musculoskeletal and connective tissue disorders) | 90 | 102
Myalgia (Musculoskeletal and connective tissue disorders) | 226 | 248
Pain in extremity (Musculoskeletal and connective tissue disorders) | 328 | 332
Dizziness (Nervous system disorders) | 150 | 145
Dysgeusia (Nervous system disorders) | 95 | 61
Headache (Nervous system disorders) | 304 | 325
Peripheral sensory neuropathy (Nervous system disorders) | 484 | 517
Anxiety (Psychiatric disorders) | 251 | 241
Depression (Psychiatric disorders) | 243 | 242
Insomnia (Psychiatric disorders) | 417 | 380
Breast pain (Reproductive system and breast disorders) | 111 | 145
Vaginal dryness (Reproductive system and breast disorders) | 99 | 99
Cough (Respiratory, thoracic and mediastinal disorders) | 159 | 171
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 165 | 170
Alopecia (Skin and subcutaneous tissue disorders) | 194 | 159
Hot flashes (Vascular disorders) | 716 | 706
Hypertension (Vascular disorders) | 207 | 227
Lymphedema (Vascular disorders) | 171 | 178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT01101438/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT01101438/SAP_001.pdf